CLINICAL TRIAL: NCT03618407
Title: Effect of Early Antiviral Therapy on Duration of Cough in Flu Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, HuKe, Director of Respiratory and Critical Care Medicine II, Renmin Hospital of Wuhan University
Other Study IDs: HuKe
Record Dates: First submitted 2018-07-04; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Influenza Virus Infection
Keywords: Influenza; Antiviral Treatment; Cough; Oseltamivir capsule; Lotus Clear Capsule
MeSH Terms: conditions — Influenza, Human; Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples Saliva samples Sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral oseltamivir group: Patients with influenza virus positive and early oral oseltamivir capsules
- Oral Lotus Capsules group: Patients with positive influenza virus and early oral administration of lotus extract capsules
- other group: Influenza virus positive patients who were not treated with oral lotus capsule or oseltamivir capsules early

SUMMARY:
This study mainly focused on the effect of early antiviral treatment on the duration of cough in influenza patients.investigators conducted an early investigation of patients with positive influenza virus and asked whether patients used antiviral drugs in the early stages. According to the use of drugs, patients were divided into oral oseltamivir group, oral lotus phlegm group and other groups, and investigators will collected Inspection information and medication status,during the treatment period of patients.

DETAILED DESCRIPTION:
Cough is a common symptom of respiratory diseases and helps to clear respiratory secretions and harmful factors, but frequent severe coughing has a serious impact on the patient's work, life and social activities. Upper respiratory tract viral infection is a common cause of coughing. Many patients have a long duration of cough after suffering from flu. Cough can last for several weeks, and most often have irritating dry cough or a small amount of white mucus sputum. This type of cough is also often referred to as "subacute cough" or "post-infection cough." The mechanisms that cause this cough have not been fully elucidated, and the effect of conventional treatment is not good, and chest imaging has no obvious abnormalities. The use of large amounts of antibiotics is ineffective or ineffective. Antihistamine H1 receptor antagonists and central antitussives are often only effective or ineffective in the short term. The effects of various bronchodilators and even hormone drugs are not clear. Due to the poor efficacy of multiple treatments, patients are repeatedly subjected to various tests, which not only increases the pain but also aggravates the economic burden.

Therefore, it is necessary to further clarify the causes and treatment measures of post-influenza cough patients.

ELIGIBILITY:
Inclusion Criteria:

For patients with flu-free flu, cough for at least one week.

1. In line with the flu etiological diagnostic criteria: According to the guidelines set by the National Health and Health Committee, the diagnosis is based on etiological screening methods or confirmed methods; ages 18 to 70 years.
2. There are no influenza complications such as acute lower respiratory tract infection, tonsillitis, sinusitis, otitis media, myocarditis, etc.
3. It is usually healthy and there are no chronic underlying diseases such as hypertension and diabetes.
4. Treating with cough as the main symptom, the cough lasts for at least one week and the chest radiograph is normal.
5. Signed informed consent.

Exclusion Criteria:

1. Suspected flu patients who have not received the flu etiology test;
2. There is a clear comorbid disease (combined with other sites of acute bacterial or viral infections);
3. There is a clear cough caused by other reasons;
4. With severe liver and kidney dysfunction;
5. Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flu patients who were diagnosed in our hospital from April 2018 to July 2019
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Cough duration | 6 months
  Investigators will follow up every other week for follow-up calls or outpatients to ask about cough and medication, until the patient stops coughing, cough lasts from 1 day to 12 weeks, and cough time is greater than 12 weeks. Investigators should seriously exclude cough caused by other factors. No other factors are still included in the study, and the maximum time is no more than 6 months. If there are other factors causing cough, it will not be included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided